CLINICAL TRIAL: NCT06224803
Title: Evaluation of Effects of Dibifree® on Regulation of Blood Sugar and HbA1c in Patients With Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Preventive Medicine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DF202006001
Record Dates: First submitted 2024-01-08; First posted 2024-01-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Baseline physical examinations were conducted at the time of inclusion (V0), including assessments of fasting and postprandial blood sugar, HbA1c, body fat, blood urea nitrogen (BUN), creatinine (CRE), estimated glomerular filtration rate (eGFR), total cholesterol, HDL-cholesterol, LDL-cholesterol, Glutamic Oxaloacetic Transaminase (GOT), and Glutamic Pyruvic Transaminase (GPT). These parameters were routinely monitored in the third month (V3), fourth month (V4), and seventh month (V7). No adjustments were made to the diabetic routine medications during the clinical trial period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dibifree (Experimental): Participants were instructed to consume ten Dibifree capsules each time, 5 to 10 minutes before meals, three times daily, for three months. This course of treatment was followed by a one-month washout period, after which Dibifree was resumed for an additional three months.
  Interventions: Dietary Supplement: Compound plant extracts
- Control (Placebo Comparator): Participants were instructed to take ten starch-containing placebo capsules 5 to 10 minutes before meals , three times daily, for three months. This was followed by a one-month washout period, after which participants switched to Dibifree treatment at the same dosage as the experimental group for another three months.
  Interventions: Dietary Supplement: Indigestible dextrin

INTERVENTIONS:
Dietary Supplement: Compound plant extracts — Total supplement including bitter melon (Momordica charantia) fruit extract, celery (Apium graveolens) seed extract, baker's yeast (Saccharomyces cerevisiae) cell wall extract, acerola (Malpighia emarginata) fruit extract, grape (Vitis vinifera) seed extract, green tea leaf extract, and hydrolyzed soy protein powder.
  Other Names: Dibifree
  Arms: Dibifree
Dietary Supplement: Indigestible dextrin — Indigestible dextrin as placebo intervention
  Other Names: Control
  Arms: Control

SUMMARY:
At present, diabetic patients mainly use drugs to control blood sugar. However, drugs have side effects and the control effect varies among individuals. Even if diabetic patients can control their blood sugar well, long-term medication will still cause a series of complications, including retinopathy, nephropathy, diabetic foot, heart disease, etc. Vascular disease issues, etc.

This study will focus on the changes in HbA1c and blood sugar in patients with confirmed diabetes after taking "Dibifree®" food supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 years old (inclusive) or above, gender is not restricted
2. Diagnosed with type 2 diabetes
3. HbA1c > 6.5%
4. Coagulation function and platelets are normal
5. Participants voluntarily join this treatment course and sign the informed consent form
6. Not taking other supplements containing blood sugar regulating properties for at least one month

Exclusion Criteria:

1. Women who are pregnant, lactating or planning to have children
2. Have factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.
3. Uncontrolled hypertension (>180/110 mmHG)
4. People suffering from stroke, elderly dementia, Alzheimer's disease and other brain diseases
5. During this study, the subject used other drugs or treatments that may interfere with this study in addition to blood sugar control medications.
6. GOT>4 times normal value; GPT>4 times normal value
7. Creatinine>4 times the highest normal value
8. Those who are determined by the project administrator to be unfit to participate in this clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Concentration of HbA1c | HbA1c was measured at baseline (V0) and during follow-up visits at months 3 (V3), 4 (V4), and 7 (V7) after intervention.
  Hemoglobin A1c (HbA1c) levels were measured at baseline (V0) and routinely monitored at the third (V3), fourth (V4), and seventh (V7) months. For longitudinal analysis, repeated measures were evaluated using two-way ANOVA followed by Sidak's multiple comparisons test to assess time and treatment effects. Data are presented as mean ± SD. All statistical analyses were performed using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA). All data were considered statistically significant at p ≤ 0.05.
Body Weight and BMI | Body weight and BMI were measured at baseline (V0) and at the end of the 7-month intervention (V7).
  Changes in body weight and BMI between baseline (V0) and month 7 (V7) were analyzed using an unpaired t-test. Statistical analyses were conducted using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA), with p ≤ 0.05 considered statistically significant.

SECONDARY OUTCOMES:
Concentration of Blood Sugar | measured at baseline (V0) and during follow-up visits at months 3 (V3), 4 (V4), and 7 (V7) after intervention.
  AC & PC blood sugar levels were measured at baseline (V0) and routinely monitored at the third (V3), fourth (V4), and seventh (V7) months. For longitudinal analysis, repeated measures were evaluated using two-way ANOVA followed by Sidak's multiple comparisons test to assess time and treatment effects. Data are presented as mean ± SD. All statistical analyses were performed using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA). All data were considered statistically significant at p ≤ 0.05.
Kidney Function Parameters: BUN, Creatinine, and eGFR | Kidney function parameters measured at baseline (V0) and during follow-up visits at months 3 (V3), 4 (V4), and 7 (V7) after intervention.
  Kidney Function Parameters were measured at baseline (V0) and routinely monitored at the third (V3), fourth (V4), and seventh (V7) months. For longitudinal analysis, repeated measures were evaluated using two-way ANOVA followed by Sidak's multiple comparisons test to assess time and treatment effects. Data are presented as mean ± SD. All statistical analyses were performed using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA). All data were considered statistically significant at p ≤ 0.05.
Liver Function Parameters: GOT and GPT | Liver function parameters measured at baseline (V0) and during follow-up visits at months 3 (V3), 4 (V4), and 7 (V7) after intervention.
  Liver Function Parameters were measured at baseline (V0) and routinely monitored at the third (V3), fourth (V4), and seventh (V7) months. For longitudinal analysis, repeated measures were evaluated using two-way ANOVA followed by Sidak's multiple comparisons test to assess time and treatment effects. Data are presented as mean ± SD. All statistical analyses were performed using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA). All data were considered statistically significant at p ≤ 0.05.
Concentration of blood lipid | The measurement at baseline (V0) and during follow-up visits at months 3 (V3), 4 (V4), and 7 (V7) after intervention.
  Total cholesterol, HDL-cholesterol, and LDL-cholesterol were measured at baseline (V0) and routinely monitored at the third (V3), fourth (V4), and seventh (V7) months. For longitudinal analysis, repeated measures were evaluated using two-way ANOVA followed by Sidak's multiple comparisons test to assess time and treatment effects. Data are presented as mean ± SD. All statistical analyses were performed using GraphPad Prism 10 (GraphPad Software, San Diego, CA, USA). All data were considered statistically significant at p ≤ 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Global Preventive Medicine Biotech Co., Ltd., New Taipei City, NEW TAIPEI, Taiwan

IPD SHARING:
Plan to Share IPD: No